CLINICAL TRIAL: NCT00203476
Title: A Prospective, Open Label Comparison of Ezetimibe, Niacin, and Colestipol as Adjunct Therapy in Lipid Reduction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tuscaloosa Research & Education Advancement Corporation (Other)
Collaborators: American Society of Health-System Pharmacists Research and Education Foundation (Other)
Responsible Party: Principal Investigator, Raela Williford, PharmD, Clinical Pharmacist/PI, Tuscaloosa Research & Education Advancement Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TREAC Cholesterol Study; TREAC Cholesterol Study
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2014-08-12 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Hyperlipidemia; Hypercholesterolemia
Keywords: ezetimibe; niacin; colestipol; hyperlipidemia; adjunct therapy; zetia
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia | interventions — Niacin; Colestipol; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Statin with Niacin (Active Comparator): Niacin dose range of 500-1500mg (average 888mg)
  Interventions: Drug: Niacin
- Statin with Colestipol (Active Comparator): Colestipol dose range 5-15gm (average 9.5gm)
  Interventions: Drug: Colestipol
- Statin with Ezitimibe (Active Comparator): Ezitimibe 10mg (average 10mg)
  Interventions: Drug: Ezetimibe

INTERVENTIONS:
Drug: Niacin
  Arms: Statin with Niacin
Drug: Colestipol
  Arms: Statin with Colestipol
Drug: Ezetimibe
  Other Names: Zetia
  Arms: Statin with Ezitimibe

SUMMARY:
To compare LDL reduction compared to baseline in patients using maximum tolerated HMG CoA Reductase inhibitor (statin) therapy with adjunctive therapy with ezetimibe, colestipol, or niacin. The patient's cardiovascular risks are assessed to determine if National Cholesterol Education Program's Adult Treatment Panel III (NCEP ATP III) guidelines for low density lipoprotein (LDL) reduction were achieved between the three groups. Secondary measures examine the safety issues with liver function test (LFT) monitoring and rhabdomyolysis. High-density lipoproteins (HDL) elevations are monitored between the three groups to determine efficacy as a secondary outcome.

DETAILED DESCRIPTION:
: Patients with hyperlipidemia who sign consent and who are currently at maximum tolerated dose of a statin and are not meeting NCEP ATPIII treatment goals for LDL cholesterol are enrolled in 12-week open label, prospective trial. Patients are randomized into one of three groups to receive ezetimibe, niacin, or colestipol in addition to current statin therapy. Patients are titrated as tolerated to therapeutic doses of study medications (ezetimibe 10mg/day, niacin 1500mg/day, and colestipol 20gm/day). At baseline, informed consent; a laboratory admission profile (Chem20); weight; height; blood pressure; concomitant medications; cholesterol medication history; and grapefruit juice consumption data are gathered. At weeks 6 and 12, patients have their cholesterol panels and liver function tests assessed. Patients are also interviewed regarding side effects (including rhabdomyolysis), tolerance, changes in concomitant medications, and grapefruit juice consumption, along with weight and blood pressure measurements.

ELIGIBILITY:
Inclusion Criteria:

* Veterans eligible for treatment at the Tuscaloosa VA Medical Center
* 50 years of age
* Male or female
* Any race or ethnic group
* Signed informed consent
* Hyperlipidemia despite current maximum tolerated dose of an HMG CoA Reductase inhibitor (statin) for > 6 weeks
* Currently not meeting NCEP ATPIII treatment goals for LDL cholesterol

Exclusion Criteria:

* Known hypersensitivity or intolerance to ezetimibe, niacin, or colestipol
* Previous failed adequate trial of adjunctive ezetimibe, niacin, or colestipol
* Consumes more than 8oz. grapefruit juice daily
* Significant medical condition that would impact safety evaluations (i.e. significantly elevated LFT, hepatitis, severe dermatitis, uncontrolled diabetes, severe GI disease, fibromyalgia, renal failure, recent CVA or MI, pancreatitis, etc.)
* Receiving medications that would be contraindicated to use in combination with ezetimibe, niacin, or colestipol

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-05; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raela B Williford, PharmD, Principal Investigator — Tuscaloosa Veterans Affairs Medical Center
Locations (1):
- Tuscaloosa Research & Education Advancement Corporation, Tuscaloosa, Alabama, United States

REFERENCES:
- [Background] Ansell BJ. Rationale for combination therapy with statin drugs in the treatment of dyslipidemia. Curr Atheroscler Rep. 2005 Feb;7(1):29-33. doi: 10.1007/s11883-005-0072-7. PMID 15683599

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 2005-2007 from primary care medical clinics.
Pre-assignment Details: Patients had to be on max tolerated dose of a statin and need additional LDL lowering.
Groups:
- Niacin: Niacin added to max tolerated dose of statin
- Colestipol: Colestipol added to max dose statin
- Ezetimibe: Ezetimibe added to max tolerated dose statin
Period: Overall Study
Arm/Group | Niacin | Colestipol | Ezetimibe
Started | 10 | 10 | 10
Completed | 9 | 9 | 10
Not Completed | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: 100% male, age 50 years or greater
Groups:
- Total: Total of all reporting groups
Arm/Group | Niacin | Colestipol | Ezetimibe | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Customized [Number; unit: participants]
  Age =>50 | 10 | 10 | 10 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 10 | 10 | 10 | 30
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: LDL Goal Attainment
Description: Each participant had his LDL goal calculated based on the NCEP ATPIII guidelines.
Time Frame: 12 weeks
Population: intention to treat
Measure: Number; unit: participants
Arm/Group | Niacin | Colestipol | Ezetimibe
Number analyzed (Participants) | 9 | 9 | 10
participants | 6 | 6 | 9

2. Secondary Outcome: LFT Elevation
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Niacin | Colestipol | Ezetimibe
Number analyzed (Participants) | 9 | 9 | 10
participants | 1 | 1 | 2

3. Secondary Outcome: Incidents of Rhabdomyolysis
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Niacin | Colestipol | Ezetimibe
Number analyzed (Participants) | 9 | 9 | 10
participants | 0 (30.55) | 0 (12.97) | 0 (20.07)

4. Secondary Outcome: Change in HDL From Baseline to 12 Weeks.
Time Frame: baseline and 12 weeks
Population: Change in HDL
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Niacin | Colestipol | Ezetimibe
Number analyzed (Participants) | 9 | 9 | 10
mg/dl
  baseline | 42.33 (11.20) | 39.22 (14.22) | 32.90 (5.15)
  12 weeks | 43.00 (11.62) | 37.56 (7.83) | 34.70 (10.39)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Niacin | Colestipol | Ezetimibe
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 6/10 | 3/10 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Niacin (N=10) | Colestipol (N=10) | Ezetimibe (N=10)
Elevated LFTs (Hepatobiliary disorders) | 1 | 1 | 2 — 1 participant in the ezetimibe group had LFTs >3 x upper limit of normal. All other elevated LFTs were not 3 x ULN.
Indestion and belching (Gastrointestinal disorders) | 0 | 0 | 1
Flushing (Skin and subcutaneous tissue disorders) | 5 | 0 | 0
Loose Stools (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Edema (Vascular disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Open label.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No